CLINICAL TRIAL: NCT06446336
Title: Creation of a Pre-operative Score, the HASS Score, for Injuries Reliable Diagnosis of Long Biceps Tendon
Acronym: HASS
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: RGDS-2023-12-010
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Biceps Tendon Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: HASS Score — Creation of a pre-operative score

SUMMARY:
The long biceps tendon (LBT) has a particular anatomical pathway, making it fragile due to repeated microtrauma or trauma which can lead to chronic lesions of LBT.

Current issue with this pathology is the absence of preoperative effective clinical and paraclinical tools, allowing confirmed diagnosis, in particular because of its entanglement with other pathologies.

This diagnostic uncertainty generates an approximation for LBT therapeutic indications so that therapeutic indications are frequently finalized during glenohumeral arthroscopy.

Having a reliable and reproducible diagnostic tool for LBT pathologies would allow an improvement in their surgical load management .

In this context, this research is based on the hypothesis that the construction of a pre-operative score, the HASS score, combining pre-operative clinical and paraclinical data would allow to obtain a reliable diagnosis of LBT injuries.

DETAILED DESCRIPTION:
The long biceps tendon (LBT) has a particular anatomical pathway, making it fragile due to repeated microtrauma or trauma which can lead to chronic lesions of LBT. Aging can also worsen damage to this tendon. LBT lesions are frequently associated with other pathologies of glenohumeral complex, particularly damage to the rotators' cuff or subacromial impingements.

Current issue with this pathology is the absence of preoperative effective clinical and paraclinical tools, allowing confirmed diagnosis, in particular because of its entanglement with other pathologies.

Isolated clinical tests are numerous and ineffective. Ultrasound is a reliable examination for taking LBT volumetric measurements or to diagnose instability but it fails in the diagnosis of cracks and tendinopathy. CT scan, CT arthrography, MRI and MRI arthrography, except a few characteristic signs of LBT lesions, ignore most of lesions and their analysis is difficult and little reproducible.

This diagnostic uncertainty generates an approximation for LBT therapeutic indications so that therapeutic indications are frequently finalized during glenohumeral arthroscopy. However, more distal lesions, in or under the bicipital groove, not accessible in arthroscopy, are described in the literature.

Having a reliable and reproducible diagnostic tool for LBT pathologies would allow an improvement in their surgical load management . It would then be possible not to ignore a lesion which is not visible on arthroscopy or conversely not to perform excess gestures on healthy LBT. It would allow also to provide clear preoperative information to patient on planned surgical procedures and their consequences.

In this context, this research is based on the hypothesis that the construction of a pre-operative score, the HASS score, combining pre-operative clinical and paraclinical data would allow to obtain a reliable diagnosis of LBT injuries.

ELIGIBILITY:
Inclusion Criteria:

* Patient with operative indication for tenodesis tenotomy, represented by persistence of clinical signs after medical treatment for more than 6 months
* Patient with shoulder pain lasting more than 6 months

Exclusion Criteria:

* Patient with a ruptured LBT on the pre-operative imaging assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who fulfill eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
HASS score | 1 day
  HASS score will rely on clinical data (Speed test, O'Brien test, palpation of the bicipital groove, Yergason test, Uppercut test, Throwing test and Hourglass test) and imaging data (Scan or CT scan, MRI or arthro-MRI)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé de l'Estuaire, Le Havre, France

IPD SHARING:
Plan to Share IPD: No